CLINICAL TRIAL: NCT05439473
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Curalin as Add-On Therapy in Adults With Type 2 Diabetes Mellitus
Brief Title: Evaluation of the Efficacy and Safety of Curalin as Add-On Therapy in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CuraLife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cura-02
Record Dates: First submitted 2021-06-08; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Type2 Diabetes
Keywords: Diabetes; Type 2 Diabetes; placebo; Curalin; CuraLife; Momordica Charantia; Gymnema Sylvestre; Trigonella Foenum Graecum; Curcuma Longa; Emblica Officinalis; Swertia Chirata; Picrorhiza Kurroa; Syzygium Cumini/ Eugenia Jambolana; Cinnamomum Zeylanicum
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Curalin
- Treatment (Active Comparator)
  Interventions: Dietary Supplement: Curalin

INTERVENTIONS:
Dietary Supplement: Curalin — Supplement capsules, 2 capsules, 3 times a day after meals. Placebo: matching placebo capsules, 2 capsules, 3 times a day after meals.

SUMMARY:
Evaluation of Efficacy and Safety of Curalin As Add-On Therapy in Adults With Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Curalin As Add-On Therapy in Adults With Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* Adult patients (18-85 years of age) with Type II diabetes mellitus.
* HbA1c at screening is 8% - 11%.
* Body mass index (BMI)>25.
* Stable body weight (±10%) within the 3 months preceding study entry.
* Patients were steadily treated with anti-diabetic medications, such as: GLP-1, Glucophage DPP-4 inhibitor or SGLT-2 inhibitor for at least 3 months or more prior to study entry.
* The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow up evaluation as specified in this protocol.

Exclusion Criteria:

* Patients who have been using Curalin
* Persons with known sensitivity to any of the components of the Curalin product.
* The patient has any clinically significant uncontrolled medical condition (treated or untreated).
* Patients with renal insufficiency (glomerular filtration rate [GFR]≤30 mL/min/1.73m2).
* Pregnant or lactating women. Women of child bearing potential will be administered a urine pregnancy test at study entry. All study participants will confirm their willingness to use birth control throughout the study.
* Patients deemed by the Investigator as unable to complete study participation.
* Patients currently treated with insulin or those that have been treated with insulin for more than 10 days in the 3 months prior to study entry.
* Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, local, dermal and inhaled steroids, and immunosuppressive or immunomodulating agents for more than a month prior to study entry, or during the study.
* Patient participated in a clinical study (investigational study drug or study device) within 30 days of the study entry.
* Life expectancy less than 1 year.
* History of stroke, transient ischemic attack, or myocardial infarction within six months prior to screening.
* Patients with uncontrolled hypertension defined as a systolic blood pressure ≥180 mmHg or a diastolic blood pressure ≥100mmHg.
* Patients who have thyroid stimulating hormone (TSH) levels >1.5 times the upper limit of normal.
* Patients with significant liver disease or liver function impairment defined as any of the following; cirrhosis, hepatitis, biliary obstruction with hyperbilirubinemia (total bilirubin >2 times the upper limit of normal) and aspartate aminotransferase (AST) or alanine aminotransferase levels (ALT) >3 times the upper limit of normal.
* Patients with creatine kinase concentrations > 10 times the upper limit of normal or creatine kinase elevation due to known muscle disease at visit 1 (screening 1).
* Laboratory abnormalities at screening including:
* Potassium > 5.5 mEq/L
* Sodium ≤ 130 mEq/L
* Hemoglobin under 10 g/dl for Women or Under 11 g/dl for man.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Effect of treatment with Curalin on the change in plasma HbA1c | 1 month
  The primary objective of this study is to evaluate the effect of treatment with Curalin on the change in plasma HbA1c.
  Glycated hemoglobin (HbA1c) is a form of hemoglobin that is measured primarily to identify the three-month average plasma glucose concentration. The primary endpoint of the study is HbA1c at 1 month.
  Blood for HbA1c will be taken at Screening, and M1/Termination of Study. HbA1c level will be ascertained at the local lab, according to the lab's operating procedures
  Rate of patients that significantly improved their HbA1c levels at least 0.5%.

SECONDARY OUTCOMES:
Effect of Curalin on Fructosamin based on blood tests | 1 month
  To evaluate the effect of Curalin on Fructosamin level based on blood tests(mmol/L)
Efect of Curalin on Fasting Blood Glucose Blood for glucose assessment | 1 month
  To evaluate the effect of Curalin on Fasting Blood Glucose Blood for glucose assessment will be taken after a 12 hour fast at Screening, Baseline, and M1/Termination of PC Study.
  Fasting blood glucose level will be ascertained at the local site lab, according to the site's operating procedures.
  In addition, participants will self-monitor their blood glucose levels at home once a week using a blood glucose meter.
Safety of Curalin as assessed by adverse events | 1 month
  To evaluate the safety of Curalin as assessed by adverse events, including the following:
  * Fasting blood chemistry including (in addition to the efficacy variables of Fructosamine): HbA1c, glucose, urea, creatinine, phosphorus, calcium, potassium, albumin, sodium (Na+) and liver function tests (ALT, AST, bilirubin and GGT), GFR, CBC.
  * Vital Signs including (in addition to the efficacy variable of blood pressure): pulse rate, body temperature

CONTACTS AND LOCATIONS:
Locations (1):
- DMC, Tel Aviv, Israel